CLINICAL TRIAL: NCT03734458
Title: Platelet Rich Fibrin and Autologous Fibrin Glue for Treating Periodontal Recession Defects: a Comparative Clinical Study
Brief Title: Platelet Rich Fibrin and Autologous Fibrin Glue
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IND application did not get approved
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-24111 PRF+AFG
Record Dates: First submitted 2018-10-03; First posted 2018-11-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - PRF plus AFG with a CAF (Experimental): Group A - PRF plus AFG with a CAF: The PRF will be prepared according to the protocol outlined by Choukroun 1. Prior to the surgical procedure, venous blood will be collected via venipuncture from the antecubital vein using one 10 ml sterile glass tube and one 10ml sterile plastic tube. The tubes will be immediately centrifuged at 1300 rpm for 8 minutes to obtain PRF. The fibrin clot formed in the middle part of the tube will be collected. The clot will be transferred to the PRF box and compressed to form a membrane. For the AFG, the liquid will be separated from the red blood cells from the plastic tube using a sterile syringe.
  Interventions: Other: Group A - PRF plus AFG with a CAF
- Group B - PRF only with a CAF (Experimental): Group B - PRF only with a CAF: The PRF will be prepared according to the protocol outlined by Choukroun1. Prior to the surgical procedure, venous blood will be collected via venipuncture from the antecubital vein using one 10 ml sterile glass tube. The tubes will be immediately centrifuged at 1300 rpm for 8 minutes to obtain PRF. The fibrin clot formed in the middle part of the tube will be collected. The clot will be transferred to the PRF box and compressed to form a membrane.
  Interventions: Other: Group B - PRF only with a CAF
- Group C - CTG with a CAF (Active Comparator): Group C - CTG with a CAF: Sup-epithelial connective tissue harvest: The palatal donor site should be at least 3mm in thickness. A horizontal incision will be made on the palate 3mm from the maxillary canine to the first molar using a 15 blade. A sub-epithelial connective tissue graft will be harvested with adequate dimensions based on the recipient site. The graft will be sutured over the recipient site with 5-0 chromic gut sutures using a continuous mattress suturing technique.
  Interventions: Other: Group C - CTG with a CAF

INTERVENTIONS:
Other: Group A - PRF plus AFG with a CAF — Group A - PRF plus AFG with a CAF will be used surgically to cover the exposed roots.
  Arms: Group A - PRF plus AFG with a CAF
Other: Group B - PRF only with a CAF — Group B - PRF only with a CAF will be used surgically to cover the exposed roots.
  Arms: Group B - PRF only with a CAF
Other: Group C - CTG with a CAF — Group C - CTG with a CAF will be used surgically to cover the exposed roots.
  Arms: Group C - CTG with a CAF

SUMMARY:
Platelet-rich fibrin (PRF) and Autologous Fibrin Glue (AFG) are fibrin preparation derived from human blood samples and are used in regenerative dentistry.

Aim: The aim of this study is to evaluate the level of root coverage using PRF (+) AFG with a coronally advanced flap (CAF) or PRF only with a CAF compared to a sub-epithelial connective tissue graft (CTG) with a CAF for treating Class 1 and 2 gingival recession defects. Additionally, to evaluate the level of keratinized tissue tissue thickness and width using PRF (+) AFG with a CAF or PRF only with a CAF compared to CTG with CAF for Class 1 and 2 gingival recession defects.

Method: 48 patients with recession defects will be randomly divided into three different treatment groups. Treatment Group A (n=16) will consist of patients treated with PRF (+) AFG with a CAF, Group B (n=16) will consist of patients treated with PRF only with a CAF and Group C (n=16) will consits of patients treated with CTG with CAF as a control. Clinical measurements will be assessed at baseline and at 1 month and 6 months after the surgery. The clinical measurements that will be recorded, include probing depth, clinical attachment level, and gingval recession parameters. The gingival recession parameters include recession width, depth and thickness.

DETAILED DESCRIPTION:
Specific aim 1: Evaluate the level of root coverage using Platelet Rich Fibrin (PRF) plus Autologous Fibrin Glue (AFG) with a coronally advanced flap (CAF) or PRF only with a CAF compared to subepithelial connective tissue graft (CTG) with a CAF for Class 1 and 2 gingival recession defects.

Specific aim 2: Evaluate the level of keratinized tissue thickness and width using PRF plus AFG with a CAF, PRF only with a CAF or a SCTG with CAF for Class 1 and 2 gingival recession defects.

Research design and methods:

Subjects and treating clinician will not be aware of the treatment arm until immediately before the surgery. Each treatment arm will use the same surgical protocol for treating gingival recession and will differ by the material used to cover the tooth root. Intervention A will use PRF with the addition of AFG. Intervention B will use PRF. The control arm will use CTG.

Methods: A total of 48 patients with recession defects will be randomly assigned to three different treatment groups. Treatment group A (n=16) will consist of patients treated with PRF plus AFG with a CAF, Group B (n=16) will consist of patients treated with PRF with a CAF and Group C (n=16) will consist of patients treated with CTG with a CAF. Group C will be the control group. Clinical measurements, including recession defect length and gingival width and thickness, will be evaluated at baseline, one month and six months after treatment. For standardization, measurements will be taken using pre- fabricated stents with an endo file stopper. A visual analogue scale will be used to compare post-operative pain between the two procedures.

Study Subjects Overview: This study will use the patient pool of the periodontal clinic at the UCSF Dental Center to identify potentially eligible patients. The periodontal clinic regularly receives a high volume of referred patients for treatment of gingival recession.

Inclusion Criteria:

1. Men and women aged 18 years or over 2. Miller's Class 1 and Class 2 recession Miller's Class 1 - Marginal tissue recession which does not extend to the mucogingival junction. There is no periodontal loss (bone or softi tssue ) in the interdental area, and 100% root coverage can be anticipated.

Miller's Class 2 - Marginal tissue recession which extends beyond the mucogingival junction.There is no periodontal loss (bone or softi tssue ) in the interdental area, and 100% root coverage can be anticipated.

5 Localized gingival recession of 1-6mm present on 1 or 2 continuous single rooted teeth. Gingival recession is measured from the cemental-enamel junction (CEJ; a stable anatomical landmark on every tooth) to the gingival margin.

Exclusion Criteria:

1. Current tobacco use (greater than 1 cigarette/week) or history of quitting < 5 years previously (self reported)
2. Poor oral hygiene (plaque index of 2 or greater) or active periodontal disease (diagnosis of moderate chronic periodontal disease or greater)
3. Currently taking aspirin, prescription blood thinners, or present with any coagulopathies 4. Type II diabetes with HbA1c greater than 7

5. Immunosuppressed or any other systemic condition that would disqualify subject as an acceptable surgical candidate Retention strategy: In the course of review if funding becomes available modest financial incentives will be made to patients returning for the 1 month and 6 month recall appointments. Otherwise, telephone and email reminders will be made by study staff for recall appointments.

PRF Preparation The PRF will be prepared according to the protocol outlined by Choukroun 1. Prior to the surgical procedure, venous blood will be collected via venipuncture from the antecubital vein using two 10 ml sterile glass tube and one 10ml sterile plastic tube. The tubes will be immediately centrifuged at 1300 rpm for 8 minutes to obtain PRF. The fibrin clot formed in the middle part of the tube will be collected. The clot will be transferred to the PRF box and compressed to form a membrane. For the AFG, the liquid will be separated from the red blood cells from the plastic tube using a sterile syringe.

Sup-epithelial connective tissue harvest:

The palatal donor site should be at least 3mm in thickness. A horizontal incision will be made on the palate 3mm from the maxillary canine to the first molar using a 15 blade. A sub-epithelial connective tissue graft will be harvested with adequate dimensions based on the recipient site. The graft will be sutured over the recipient site with 5-0 chromic gut sutures using a continuous mattress suturing technique.

Surgical procedure:

An acrylic stent will be made using patient's models/dental cast. On the day of the procedure, the recession defect length and width will be measured using the pre-fabricated stent and periodontal probe. The gingival thickness will be evaluated using an endo reamer and stopper. For all groups, the recipient bed will be prepared using a horizontal sulcular incision. A split thickness flap will be reflected to expose the periosteum. The flap will be extended mesio-distally from the recession defect for adequate blood supply and for passive primary closure. For Group C - CTG w/ CAF, the CTG harvested from the palate will be placed over the recession defect. For Group B PRF w/CAF, the PRF membrane will be placed on the recession defect. For Group A -PRF plus AFG w/ CAF, the AFG liquid will be applied over the exposed roots of the recession defect and the PRF membrane will be placed on the recession defect. For all groups, the recipient flap will cover the graft and be coronally positioned over the cemento-enamel junction. The recipient site will be sutured using a sling suturing technique with 5-0 vicryl sutures. Care will be taken to achieve tension free primary closure for all the groups. Hemostasis will be achieved by applying gentle finger pressure for up to 5 minutes.

Data collection and Analysis:

Clinical measurements will be assessed at baseline and at 1 month and 6 months after surgery. The clinical measurements will be recorded using a pre- fabricated stent and periodontal probe. The clinical measurements that will be recorded, include probing depth, clinical attachment level, and gingival recession parameters. The gingival recession parameters include recession width, depth and thickness. Presence of plaque and gingival inflammation will also be recorded using Loe & Silness Plaque and Gingival Index.

Standard clinical care:

- Each subject receives regular care for the root coverage procedure.

In brief, the regular care involves the following:

- Root coverage procedure involves coverage of the exposed root to improve esthetics, decrease caries risk and increase keratinized tissue. There are several techniques supported in the literature including the techniques used for treatment arm (Group B and Group C) of the study described below.

Study Procedures - After successful enrollment and randomization into a given treatment arm, subject are treated according to normal clinical care for the treating the soft tissue recession. Particpant's study models are taken and stent is created using the model.

The following study interventions are performed during the regular care phase:

Baseline measurement- The clinical measurements will be taken non-invasively using a pre- fabricated stent, periodontal probe and endo reamer with stopper before the surgery (baseline) and at 1 month, 6 months post surgery.

- Measurements will be recorded by the study coordinator on a coded data collection sheet. Soft tissue recession treatment groups : Group A - PRF plus AFG with a CAF - The PRF will be prepared according to the protocol outlined by Choukroun 1. Prior to the surgical procedure, venous blood will be collected via venipuncture from the antecubital vein using two 10 ml sterile glass tube and one 10ml sterile plastic tube. The tubes will be immediately centrifuged at 1300 rpm for 8 minutes to obtain PRF. The fibrin clot formed in the middle part of the tube will be collected. The clot will be transferred to the PRF box and compressed to form a membrane. For the AFG, the liquid will be separated from the red blood cells from the plastic tube using a sterile syringe.

Group B - PRF only with a CAF - The PRF will be prepared according to the protocol outlined by Choukroun1. Prior to the surgical procedure, venous blood will be collected via venipuncture from the antecubital vein using two 10 ml sterile glass tube. The tubes will be immediately centrifuged at 1300 rpm for 8 minutes to obtain PRF. The fibrin clot formed in the middle part of the tube will be collected. The clot will be transferred to the PRF box and compressed to form a membrane.

Group C - CTG with a CAF (Control) - Sup-epithelial connective tissue harvest: The palatal donor site should be at least 3mm in thickness. A horizontal incision will be made on the palate 3mm from the maxillary canine to the first molar using a 15 blade. A sub-epithelial connective tissue graft will be harvested with adequate dimensions based on the recipient site. The graft will be sutured over the recipient site with 5-0 chromic gut sutures using a continuous mattress suturing technique.

Surgical procedure:

An acrylic stent will be made using patient's models/dental cast. On the day of the procedure, the recession defect length and width will be measured using the pre-fabricated stent and periodontal probe. The gingival thickness will be evaluated using an endo reamer and stopper. For all groups, the recipient bed will be prepared using a horizontal sulcular incision. A split thickness flap will be reflected to expose the periosteum. The flap will be extended mesio-distally from the recession defect for adequate blood supply and for passive primary closure. For Group C - CTG w/ CAF, the CTG harvested from the palate will be placed over the recession defect as described above. For Group B PRF w/CAF, the PRF membrane will be placed on the recession defect. For Group A -PRF plus AFG w/ CAF, the AFG liquid will be applied over the exposed roots of the recession defect and the PRF membrane will be placed on the recession defect. For all groups, the recipient flap will cover the graft and be coronally positioned over the cemento-enamel junction. The recipient site will be sutured using a sling suturing technique with 5-0 vicryl sutures. Care will be taken to achieve tension free primary closure for all the groups. Hemostasis will be achieved by applying gentle finger pressure for up to 5 minutes.

Post operative visit (Week 1): Treated site checked for healing and oral hygiene instructions will be reviewed with the patient.

Post operative visit (Week 2): Treated site checked for healing and oral hygiene instructions will be reviewed with the patient.

Post operative visit (1 months): Treated site checked for healing and oral hygiene instructions will be reviewed with the patient. Topical local anesthetic will be applied on the treated area and the clinical measurements will be taken non-invasively using the pre-fabricated stent, periodontal probe and endo reamer with stopper at one month post surgery.

Post operative visit (6months): Treated site checked for healing and oral hygiene instructions will be reviewed with the patient. Clinical measurements are repeated as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years or over
2. Miller's Class 1 and Class 2 recession
3. Localized gingival recession of 1-6mm present on 1 or 2 continuous single rooted teeth. Gingival recession is measured from the cemental-enamel junction (CEJ; a stable anatomical landmark on every tooth) to the gingival margin.

Exclusion Criteria:

1. Current tobacco use (greater than 1 cigarette/week) or history of quitting < 5 years previously (self reported)
2. Poor oral hygiene (plaque index of 2 or greater) or active periodontal disease (diagnosis of moderate chronic periodontal disease or greater)
3. Currently taking aspirin, prescription blood thinners
4. Type II diabetes with HbA1c greater than 7
5. Immunosuppressed or any other systemic condition that would disqualify subject as an acceptable surgical candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18years and over.
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the level of root coverage using PRF plus AFG with a coronally advanced flap or PRF only with a CAF compared to subepithelial connective tissue graft with a CAF for Class 1 and 2 gingival recession defects. | Baseline to 6 months
  To evaluate the level of root coverage using PRF plus AFG compared to CTG or PRF only compared to CTG

SECONDARY OUTCOMES:
Evaluate the level of keratinized tissue thickness and width using PRF plus AFG with a CAF, PRF only with a CAF or a SCTG with CAF for Class 1 and 2 gingival recession defects. | Baseline to 6 months
  To evaluate the level of keratinized tissue thickness and width using PRF plus AFG compared to CTG or PRF only compared to CTG

CONTACTS AND LOCATIONS:
Overall Officials: Yogalakshmi Rajendran, BDS MS, Principal Investigator — UCSF School of Dentistry
Locations (1):
- UCSF School of Dentistry, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Choukroun J, Ghanaati S. Reduction of relative centrifugation force within injectable platelet-rich-fibrin (PRF) concentrates advances patients' own inflammatory cells, platelets and growth factors: the first introduction to the low speed centrifugation concept. Eur J Trauma Emerg Surg. 2018 Feb;44(1):87-95. doi: 10.1007/s00068-017-0767-9. Epub 2017 Mar 10. PMID 28283682
- [Result] Miron RJ, Zucchelli G, Pikos MA, Salama M, Lee S, Guillemette V, Fujioka-Kobayashi M, Bishara M, Zhang Y, Wang HL, Chandad F, Nacopoulos C, Simonpieri A, Aalam AA, Felice P, Sammartino G, Ghanaati S, Hernandez MA, Choukroun J. Use of platelet-rich fibrin in regenerative dentistry: a systematic review. Clin Oral Investig. 2017 Jul;21(6):1913-1927. doi: 10.1007/s00784-017-2133-z. Epub 2017 May 27. PMID 28551729
- [Result] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687
- [Result] Dohan Ehrenfest DM, Bielecki T, Jimbo R, Barbe G, Del Corso M, Inchingolo F, Sammartino G. Do the fibrin architecture and leukocyte content influence the growth factor release of platelet concentrates? An evidence-based answer comparing a pure platelet-rich plasma (P-PRP) gel and a leukocyte- and platelet-rich fibrin (L-PRF). Curr Pharm Biotechnol. 2012 Jun;13(7):1145-52. doi: 10.2174/138920112800624382. PMID 21740377
- [Result] Oncu E. The Use of Platelet-Rich Fibrin Versus Subepithelial Connective Tissue Graft in Treatment of Multiple Gingival Recessions: A Randomized Clinical Trial. Int J Periodontics Restorative Dent. 2017 Mar/Apr;37(2):265-271. doi: 10.11607/prd.2741. PMID 28196169
- [Result] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part II: platelet-related biologic features. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e45-50. doi: 10.1016/j.tripleo.2005.07.009. Epub 2006 Jan 10. PMID 16504850
- [Result] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part III: leucocyte activation: a new feature for platelet concentrates? Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e51-5. doi: 10.1016/j.tripleo.2005.07.010. PMID 16504851
- [Result] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849
- [Result] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Result] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part V: histologic evaluations of PRF effects on bone allograft maturation in sinus lift. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):299-303. doi: 10.1016/j.tripleo.2005.07.012. PMID 16504861